CLINICAL TRIAL: NCT04376788
Title: Exchange Transfusion Versus Plasma From Convalescent Patients With Methylene Blue in Patients With COVID-19
Acronym: COVID-19
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed Mahmoud Moussa, Professor Of Internal Medicine and Hematology -BMT, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FMASU P22/2020
Record Dates: First submitted 2020-05-01; First posted 2020-05-06 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: COVID-19
Keywords: COVID-19; Exchange transfusion; Methylene blue
MeSH Terms: conditions — COVID-19 | interventions — Methylene Blue

STUDY DESIGN:
Intervention Model Description: Group I:
  Will receive exchange transfusion by venesection of 500cc blood with good replacement of one unit packed washed RBCs daily for 3 days according to daily clinical and investigational follow up
  Group II Will receive IV methylene blue 1 mg/kg IV over 30 minutes with 200 CC plasma from convalescent matching single patient by plasma extractor machine for 3 days according to daily clinical and investigational follow up.
  Group III Will receive exchange transfusion by venesection of 500cc blood with good replacement of one unit packed washed RBCs and IV methylene blue 1 mg/kg IV over 30 minutes with 200 CC plasma from convalescent matching single patient by plasma extractor machine for 3 days according to daily clinical and investigational follow up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exchange transfusion (Experimental): Will receive exchange transfusion by venesection of 500cc blood with good replacement of one unit packed washed RBCs daily for 3 days according to daily clinical and investigational follow up
  Interventions: Biological: exchange blood transfusion from normal donor
- Methylene blue with plasma (Experimental): Will receive IV methylene blue 1 mg/kg IV over 30 minutes with 200 CC plasma from convalescent matching single patient by plasma extractor machine for 3 days according to daily clinical and investigational follow up.
  Interventions: Biological: plasma from convalescent patients with COVID-19; Drug: Methylene Blue 5 MG/ML
- Exchange transfusion and methylene blue with plasma (Experimental): Will receive exchange transfusion by venesection of 500cc blood with good replacement of one unit packed washed RBCs and IV methylene blue 1 mg/kg IV over 30 minutes with 200 CC plasma from convalescent matching single patient by plasma extractor machine for 3 days according to daily clinical and investigational follow up.
  Interventions: Biological: exchange blood transfusion from normal donor; Biological: plasma from convalescent patients with COVID-19; Drug: Methylene Blue 5 MG/ML

INTERVENTIONS:
Biological: exchange blood transfusion from normal donor — IV method
  Arms: Exchange transfusion; Exchange transfusion and methylene blue with plasma
Biological: plasma from convalescent patients with COVID-19 — IV method
  Arms: Exchange transfusion and methylene blue with plasma; Methylene blue with plasma
Drug: Methylene Blue 5 MG/ML — IV method
  Arms: Exchange transfusion and methylene blue with plasma; Methylene blue with plasma

SUMMARY:
The aim of this project is to introduce way for treatment of patients with severe COVID-19 disease with respiratory complications.

DETAILED DESCRIPTION:
Study Tools AND/ OR procedure

The patients were subjected to the following:

Clinical parameters:

Complete history taking and thorough clinical examination

1. Laboratory parameters:
2. CBC with differential counts.
3. Reticulocytic count.
4. Blood film for shistocytes.
5. Serum ferritin and transferrin saturation.
6. D dimer.
7. Liver function tests, kidney function tests, electrolytes.
8. ESR.
9. CRP.
10. LDH.
11. Viral markers (HCV Ab, HBsV AG, HIV Ab).
12. ADAM'S 13 assays.
13. Serum soluble CD 25.

Other investigations:

1. Chest X ray.
2. Pelviabdominal US.
3. CT chest.
4. ECG.
5. Echocardiography

The patients will be divided into three groups, each group formed of 5 patients with severe COVID-19 or on mechanical ventilator receiving standard of care All the groups matched regarding age, sex and the severity of the disease.

Group I:

Will receive exchange transfusion by venesection of 500cc blood with good replacement of one unit packed washed RBCs daily for 3 days according to daily clinical and investigational follow up

Group II Will receive IV methylene blue 1 mg/kg IV over 30 minutes with 200 CC plasma from convalescent matching single patient by plasma extractor machine for 3 days according to daily clinical and investigational follow up.

Group III Will receive exchange transfusion by venesection of 500cc blood with good replacement of one unit packed washed RBCs and IV methylene blue 1 mg/kg IV over 30 minutes with 200 CC plasma from convalescent matching single patient by plasma extractor machine for 3 days according to daily clinical and investigational follow up.

N.B.: Convalescent plasma and regular blood will be taken from ministry of health after administrative approval All groups will receive

1. Low dose anticoagulant (LMWH 1 mg/kg/day).
2. Steroid (methyl prednisone 1 mg/ kg IV daily and according to patients' condition and presence of complications like hemophagocytosis).
3. All allergic precautions if needed like antihistaminics , epinephrine and steroid.

Close monitoring for:

1. Allergic reactions.
2. ECG changes daily.
3. Volume overload.
4. Complications of other comorbidities like DM or HTN.
5. Liver function and kidney function and organ dysfunction daily.

Terms of discontinuation:

Deterioration of clinical condition or organ functions.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients are 18 years old or above.
2. Inpatients diagnosed as severe COVID - 19 disease according to WHO criteria.
3. CT chest with extensive lung disease (ground-glass and consolidative pulmonary opacities).
4. O2 saturation less than 93% resting.
5. Respiratory rate equal or more than 30 per minute.

Exclusion Criteria:

1. Patients with pregnancy and lactation.
2. Renal failure and heart failure.
3. Contraindication for plasma or blood transfusion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-05-20 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
improvement of condition | three to five days days
  improvement of general condition of the patients as the ventilator parameters and serum level of ferritin , D dimer, CBC, oxygen level in blood and patient o2 saturation

SECONDARY OUTCOMES:
change in organs function with PFS and OS | 0ne month
  change in the liver , kidney function and change in ferritin level with normal D Dimer

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed M Moussa, MD, Principal Investigator — Ain Shams University; Ayman I Tharwat, MD, Study Director — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chang D, Lin M, Wei L, Xie L, Zhu G, Dela Cruz CS, Sharma L. Epidemiologic and Clinical Characteristics of Novel Coronavirus Infections Involving 13 Patients Outside Wuhan, China. JAMA. 2020 Mar 17;323(11):1092-1093. doi: 10.1001/jama.2020.1623. PMID 32031568
- [Background] Rothe C, Schunk M, Sothmann P, Bretzel G, Froeschl G, Wallrauch C, Zimmer T, Thiel V, Janke C, Guggemos W, Seilmaier M, Drosten C, Vollmar P, Zwirglmaier K, Zange S, Wolfel R, Hoelscher M. Transmission of 2019-nCoV Infection from an Asymptomatic Contact in Germany. N Engl J Med. 2020 Mar 5;382(10):970-971. doi: 10.1056/NEJMc2001468. Epub 2020 Jan 30. No abstract available. PMID 32003551